CLINICAL TRIAL: NCT01132508
Title: Use of a Reinforced Injectable Calcium Phosphate Bone Cement in the Treatment of Tibial Plateau Fractures
Status: Completed | Type: Observational
Sponsor: Synthes GmbH (Industry)
Collaborators: Synthes Asia Pacific (Industry)
Responsible Party: Sponsor
Other Study IDs: ND-AUS-01
Record Dates: First submitted 2010-02-16; First posted 2010-05-28 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Tibial Fractures
Keywords: Tibial plateau fracture; Orthopaedic Trauma Association (OTA) B2 B3 C3; Bone Void
MeSH Terms: conditions — Tibial Fractures; Tibial Plateau Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment
  Interventions: Device: Norian Drillable Bone Void Filler

INTERVENTIONS:
Device: Norian Drillable Bone Void Filler — Norian Drillable Bone Void Filler is a moldable, biocompatible bone void filler with added reinforcing fibers. Norian Drillable is intended to be placed into bony voids either before or after final fixation. The material can be drilled and tapped, and screws can be placed through it at any time during the setting process. Norian Drillable is a composite, two-component, self-setting calcium phosphate bone void filler
  Other Names: Norian Drillable

SUMMARY:
Case series of tibial plateau fractures using Norian Drillable.

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized prospective case series of tibial plateau fractures using Norian Drillable to fill bone voids, to evaluate OR time, blood loss, complications, ease of use, fracture stabilization and patient function and pain over time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with closed tibial plateau fractures classified as OTA B2, B3 or C3 resulting in a bone void.
* At least 18 years of age.
* Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms.
* Signed informed consent.

Exclusion Criteria:

* Critically ill
* Mentally ill or mentally disordered
* Wards of the state
* Prisoners
* Refugees
* In an employer - employee, teacher - student relationship or any other dependant with the researchers or their associates
* Active or suspected infection - systemic or local
* Gustillo classification of 2 or 3
* Bilateral tibial plateau fractures when both fracture patterns extend into the joint
* Have an existing calcium metabolism disorder (e.g. hypercalcemia)
* Chronic renal disease/renal failure
* Insulin dependent diabetes
* Taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids).
* Rheumatoid arthritis or other autoimmune disease.
* Systemic disease including AIDS, HIV, hepatitis.
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years.
* Subjects involved in other studies within the last month, prior to screening.
* Pregnant or interested in becoming pregnant in the next 18 months. Females of child-bearing potential must use an acceptable method of contraception during trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Balogh, MD, Principal Investigator — John Hunter Hospital, New Lambton, NSW, Australia; Ian Harris, MD, Principal Investigator — Liverpool Hospital, Liverpool, NSW, Australia
Locations (6):
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
- Queen Mary Hospital, Hong Kong, China
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - St. Elisabeth Ziekenhuis, Tilburg
- Sykehuset I Vestfold, Tønsberg, Norway

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 33
Treated at Baseline | 33
6 Weeks | 33
12 Weeks | 33
26 Weeks | 33
52 Weeks | 30
78 Weeks | 28
104 Weeks | 27
Completed | 24
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: All patients enrolled and treated with Norian Drillable Bone Void Filler.
Arm/Group | Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28
  Asian | 1
  Black | 0
  Indian | 0
  Other | 4
Region of Enrollment [Number; unit: participants]
  Australia | 10
  Netherlands | 6
  Norway | 16
  China | 1
Height (n=32) [Mean (Standard Deviation); unit: centimeter] | 169.5 (9.85)
Weight (n=32) [Mean (Standard Deviation); unit: kilogram] | 75.5 (18.33)
BMI (n=32) [Mean (Standard Deviation); unit: kg/m2] | 26.3 (5.78)
Exercise per week [Number; unit: participants]
  Never | 4
  1-2 times per week | 9
  3-4 times per week | 9
  5 or more times per week | 9
  Missing | 2
Occupation [Number; unit: participants]
  Retired | 12
  Student | 0
  Home worker | 2
  Office worker | 1
  Light industrial or light industrial labor | 3
  Moderate industrial or moderate physical labor | 6
  Heavy industrial or heavy industrial labor | 0
  Other | 9
Health status [Number; unit: participants]
  Excellent | 5
  Good | 18
  Fair | 9
  Poor | 0
  Missing | 1
Smoking status [Number; unit: participants]
  Never | 11
  Former | 11
  Current | 10
  Missing | 1
Injury characteristics: side of fracture [Number; unit: participants]
  Right knee | 9
  Left knee | 24
Mechanism of injury [Number; unit: participants] — Patients may had an injury in more than one category.
  participants
    Low impact trauma | 29
    High impact trauma | 7
    Sports | 6
Orthopaedic Trauma Association (OTA) fracture type [Number; unit: participants] — OTA = orthopaedic trauma association B2 = partial articular fracture classified as pure depression B3 = partial articular fracture classified as split depression C3 = complete articular fracture classified as multifragmentary
  participants
    B2 | 5
    B3 | 19
    C3 | 8
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Time the Patient Was in the OR as a Measure of Effectiveness of the Treatment
Description: Immediately after the surgery in which Norian Drillable was implanted, the surgeon completed a questionnaire in which he recorded the duration of time the patient was in the operating room (OR)
Time Frame: Day 0 (Day of surgery)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Treatment
Number analyzed (Participants) | 33
Minutes | 107.0 [52 to 392]

2. Primary Outcome: Estimate of Blood Loss in Cubic Centimeter as a Measure of Effectiveness of the Treatment
Description: Immediately after the surgery in which Norian Drillable was implanted, the surgeon completed a questionnaire in which he recorded the estimated amount of blood loss (the amount of fluid used in irrigation should have been subtracted from the amount of fluid present in the suction canister at the completion of surgery. Any gauze used in the procedure should have been estimated for the ml of blood loss)
Time Frame: Day 0 (Day of surgery)
Measure: Mean (Standard Deviation); unit: Cubic Centimeters
Arm/Group | Treatment
Number analyzed (Participants) | 31
Cubic Centimeters | 114.0 (117.35)

3. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability of the Device
Time Frame: At enrolment (between day -7 and day 0), day 0 (day of surgery), 6 weeks, 12 weeks, 26 weeks, 52 weeks, 78 weeks and 104 (for Australian sites only) postoperative
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 33
participants | 21

4. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Drill
Description: Right after the surgery in which Norian Drillable was implanted, surgeons were required to answer three questions about the ease of use of Norian Drillable.
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Easy | 27
  Moderate | 1
  Difficult | 0
  n/a | 5

5. Secondary Outcome: Pain and Function Assessed With the Lysholm Knee Scale
Description: The Lysholm Knee Score assessed pain and function of the knee (by evaluating whether support for weight bearing was needed, the patients ability to climb stairs and to squat, whether the patients knee was instable and the patient experienced pain and swelling) and was completed by the patient before surgery and at Week 6, Week 12, Week 26, Week 52, Week 78 and Week 104 (for Australian sites only). The score ranged from 0 to 100 points with higher values indicating a better healing status of the knee.
Time Frame: 6 weeks, 12 weeks, 26 weeks, 52 weeks, 78 weeks and 104 weeks (for Australian sites only)
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 28
units on a scale
  Week 6, n=24 | 52.0 [0.0 to 86.7]
  Week 12, n=23 | 66.7 [20.5 to 92.0]
  Week 26, n=20 | 70.6 [17.5 to 86.1]
  Week 52, n=24 | 75.0 [21.0 to 95.0]
  Week 78, n=21 | 67.8 [20.5 to 92.0]
  Week 104, n=4 | 73.5 [61.0 to 95.0]

6. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: K-wire
Description: Right after the surgery in which Norian Drillable was implanted, surgeons were required to answer three questions about the ease of use of Norian Drillable.
  Kirschner wires or K-wires are sterilized, sharpened, smooth stainless steel pins widely used to hold bone fragments together (pin fixation) or to provide an anchor for skeletal traction in fractures.
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Easy | 5
  Moderate | 0
  Difficult | 0
  n/a | 28

7. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Tap
Description: Right after the surgery in which Norian Drillable was implanted, surgeons were required to answer three questions about the ease of use of Norian Drillable.
  A tap is an instrument used to create threads in a hole drilled in bone.
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Easy | 8
  Moderate | 0
  Difficult | 0
  n/a | 25

8. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Screw Insertion
Description: as for outcome 4
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Easy | 29
  Moderate | 1
  Difficult | 0
  n/a | 3

9. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Product Characteristics Mixing
Description: Right after the surgery in which Norian Drillable was implanted, surgeons were required to answer five questions about the product characteristics of Norian Drillable.
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Exceptional | 6
  Very easy | 16
  Somewhat easy | 3
  Average | 6
  Fair | 1
  Somewhat difficult | 0
  Very difficult | 0
  Missing | 1

10. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Product Characteristics Handling
Description: as for outcome 9
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Exceptional | 4
  Very easy | 15
  Somewhat easy | 6
  Average | 7
  Fair | 0
  Somewhat difficult | 0
  Very difficult | 0
  Missing | 1

11. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Product Characteristics Flow Properties
Description: as for outcome 9
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Exceptional | 6
  Very easy | 9
  Somewhat easy | 10
  Average | 6
  Fair | 0
  Somewhat difficult | 1
  Very difficult | 0
  Missing | 1

12. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Product Characteristics Flexibility With Surgical Procedure
Description: as for outcome 9
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Exceptional | 2
  Very easy | 15
  Somewhat easy | 6
  Average | 9
  Fair | 0
  Somewhat difficult | 0
  Very difficult | 0
  Missing | 1

13. Primary Outcome: Ease of Use Score Measured With a Surgeon Questionnaire: Product Characteristics Overall Ease of Use
Description: as for outcome 9
Time Frame: Day 0 (Date of surgery)
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Exceptional | 6
  Very easy | 11
  Somewhat easy | 10
  Average | 4
  Fair | 0
  Somewhat difficult | 1
  Very difficult | 0
  Missing | 1

14. Secondary Outcome: Radiographic Parameters: Depression at Baseline
Description: The anatomical grading parameter "depression" was assessed the following way: Anterior-Posterior (AP) and lateral radiographs were taken for the fractured and healthy tibia plateau at Baseline, right after surgery and all follow-up timepoint. Additional oblique radiographs at 45° or other fracture imaging was optional. All post-operative radiographs were compared against the healthy tibia films post-surgery and all follow-up radiographs were compared with the post-operative radiographs to evaluate the quality and changes in reduction at each timepoint. CT scans were only mandatory at Baseline.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 0
  Present | 27
  Missing | 1

15. Secondary Outcome: Radiographic Parameters: Depression at Surgery
Description: The anatomical grading parameter "depression" was assessed the following way: AP and lateral radiographs were taken for the fractured and healthy tibia plateau at Baseline, right after surgery and all follow-up timepoint. Additional oblique radiographs at 45° or other fracture imaging was optional. All post-operative radiographs were compared against the healthy tibia films post-surgery and all follow-up radiographs were compared with the post-operative radiographs to evaluate the quality and changes in reduction at each timepoint. CT scans were only mandatory at Baseline.
Time Frame: Surgery
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 15
  Present | 12
  Missing | 1

16. Secondary Outcome: Radiographic Parameters: Depression at 6 Weeks
Description: as for outcome 15
Time Frame: 6 week
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 22
  Present | 4
  Missing | 2

17. Secondary Outcome: Radiographic Parameters: Depression at 12 Weeks
Description: as for outcome 15
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 16
  Present | 7
  Missing | 5

18. Secondary Outcome: Radiographic Parameters: Depression at 26 Weeks
Description: as for outcome 15
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 16
  Present | 5
  Missing | 7

19. Secondary Outcome: Radiographic Parameters:: Depression at 52 Weeks
Description: as for outcome 15
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 12
  Present | 8
  Missing | 8

20. Secondary Outcome: Radiographic Parameters: Depression at 78 Weeks
Description: as for outcome 15
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 13
  Present | 8
  Missing | 7

21. Secondary Outcome: Radiographic Parameters: Condylar Widening at Baseline
Description: The anatomical grading parameter "condylar widening" (enlargement of the knee joint) was assessed the following way: AP and lateral radiographs were taken for the fractured and healthy tibia plateau at Baseline, right after surgery and all follow-up timepoints. Additional oblique radiographs at 45° or other fracture imaging was optional. All post-operative radiographs were compared against the healthy tibia films post-surgery and all follow-up radiographs were compared with the post-operative radiographs to evaluate the quality and changes in reduction at each timepoint. CT scans were only mandatory at Baseline.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 6
  Present | 21
  Missing | 1

22. Secondary Outcome: Radiographic Parameters: Condylar Widening at Surgery
Description: as for outcome 21
Time Frame: Surgery
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 20
  Present | 7
  Missing | 1

23. Secondary Outcome: Radiographic Parameters: Condylar Widening at 6 Weeks
Description: as for outcome 21
Time Frame: 6 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 24
  Present | 2
  Missing | 2

24. Secondary Outcome: Radiographic Parameters: Condylar Widening at 12 Weeks
Description: as for outcome 21
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 23
  Present | 0
  Missing | 5

25. Secondary Outcome: Radiographic Parameters: Condylar Widening at 26 Weeks
Description: as for outcome 21
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 20
  Present | 1
  Missing | 7

26. Secondary Outcome: Radiographic Parameters: Condylar Widening at 52 Weeks
Description: as for outcome 21
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 20
  Present | 0
  Missing | 8

27. Secondary Outcome: Radiographic Parameters: Condylar Widening at 78 Weeks
Description: as for outcome 21
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 20
  Present | 0
  Missing | 8

28. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at Baseline
Description: The anatomical grading parameter "angulation (valgus/varus)" (abnormal outward/inward turning of the knee) was assessed the following way: AP and lateral radiographs were taken for the fractured and healthy tibia plateau at Baseline, right after surgery and all follow-up timepoints. Additional oblique radiographs at 45° or other fracture imaging was optional. All post-operative radiographs were compared against the healthy tibia films post-surgery and all follow-up radiographs were compared with the post-operative radiographs to evaluate the quality and changes in reduction at each timepoint. CT scans were only mandatory at Baseline.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 16
  Present | 9
  Missing | 3

29. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at Surgery
Description: as for outcome 28
Time Frame: Surgery
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 23
  Present | 4
  Missing | 1

30. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at 6 Weeks
Description: as for outcome 28
Time Frame: 6 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 24
  Present | 2
  Missing | 2

31. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at 12 Weeks
Description: as for outcome 28
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 21
  Present | 3
  Missing | 4

32. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at 26 Weeks
Description: as for outcome 28
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 19
  Present | 2
  Missing | 7

33. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at 52 Weeks
Description: as for outcome 28
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 17
  Present | 3
  Missing | 8

34. Secondary Outcome: Radiographic Parameters: Angulation (Valgus/Varus) at 78 Weeks
Description: as for outcome 28
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Not present | 17
  Present | 3
  Missing | 8

35. Secondary Outcome: Knee Function and Stability: Extension at Baseline
Description: The extension ability of the knee was investigated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 16
  0-10 Degrees | 10
  Missing | 2

36. Secondary Outcome: Knee Function and Stability: Extension at 6 Weeks
Description: as for outcome 35
Time Frame: 6 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 20
  0-10 Degrees | 6
  Missing | 2

37. Secondary Outcome: Knee Function and Stability: Extension at 12 Weeks
Description: as for outcome 35
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 21
  0-10 degrees | 2
  Missing | 5

38. Secondary Outcome: Knee Function and Stability: Extension at 26 Week
Description: as for outcome 35
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 18
  0-10 degrees | 3
  Missing | 7

39. Secondary Outcome: Knee Function and Stability: Extension at 52 Weeks
Description: as for outcome 35
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 20
  0-10 degrees | 4
  Missing | 4

40. Secondary Outcome: Knee Function and Stability: Extension at 78 Weeks
Description: as for outcome 35
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal | 19
  0-10 Degrees | 2
  Missing | 7

41. Secondary Outcome: Knee Function and Stability: Total Range of Motion at Baseline
Description: Total range of motion of the knee was investigated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 3
  At least 120 degrees | 4
  At least 90 degrees | 8
  At least 60 degrees | 5
  At least 30 degrees | 1
  At least 0-30 degrees | 3
  Missing | 4

42. Secondary Outcome: Knee Function and Stability: Total Range of Motion at 6 Weeks
Description: as for outcome 41
Time Frame: 6 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 4
  At least 120 degrees | 6
  At least 90 degrees | 13
  At least 60 degrees | 2
  At least 30 degrees | 2
  At least 0-30 degrees | 0
  Missing | 1

43. Secondary Outcome: Knee Function and Stability: Total Range of Motion at 12 Weeks
Description: as for outcome 41
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 10
  At least 120 degrees | 9
  At least 90 degrees | 2
  At least 60 degrees | 0
  At least 30 degrees | 2
  At least 0-30 degrees | 0
  Missing | 5

44. Secondary Outcome: Knee Function and Stability: Total Range of Motion at 26 Weeks
Description: as for outcome 41
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 4
  At least 120 degrees | 11
  At least 90 degrees | 4
  At least 60 degrees | 1
  At least 30 degrees | 1
  At least 0-30 degrees | 0
  Missing | 7

45. Secondary Outcome: Knee Function and Stability: Total Range of Motion at 52 Weeks
Description: as for outcome 41
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 16
  At least 120 degrees | 5
  At least 90 degrees | 1
  At least 60 degrees | 1
  At least 30 degrees | 1
  At least 0-30 degrees | 0
  Missing | 4

46. Primary Outcome: Surgeons Overall Satisfaction With Norian Drillable
Description: The overall satisfaction of the ease of use of Norian Drillable was rated by the surgeon.
Time Frame: Surgery
Measure: Number; unit: Cases
Arm/Group | Treatment
Number analyzed (Participants) | 33
Cases
  Very satisfied | 21
  Satisfied | 2
  Somewhat satisfied | 6
  Average | 1
  Not dissatisfied | 0
  Somewhat dissatisfied | 2
  Very dissatisfied | 0
  Missing | 1

47. Secondary Outcome: Knee Function and Stability: Total Range of Motion at 78 Weeks
Description: as for outcome 41
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  At least 140 degrees | 10
  At least 120 degrees | 9
  At least 90 degrees | 0
  At least 60 degrees | 2
  At least 30 degrees | 0
  At least 0-30 degrees | 0
  Missing | 7

48. Secondary Outcome: Knee Function and Stability: Extension Stability at Baseline
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: Baseline
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 13
  Abnormal instability | 6
  Instability in extension <10 degrees | 3
  Instability in extension >10 degrees | 1
  Missing | 5

49. Secondary Outcome: Knee Function and Stability: Extension Stability at 6 Weeks
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: 6 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 23
  Abnormal instability | 3
  Instability in extension <10 degrees | 1
  Instability in extension >10 degrees | 0
  Missing | 1

50. Secondary Outcome: Knee Function and Stability: Extension Stability at 12 Weeks
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: 12 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 22
  Abnormal instability | 1
  Instability in extension <10 degrees | 0
  Instability in extension >10 degrees | 0
  Missing | 5

51. Secondary Outcome: Knee Function and Stability: Extension Stability at 26 Weeks
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: 26 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 20
  Abnormal instability | 0
  Instability in extension <10 degrees | 1
  Instability in extension >10 degrees | 0
  Missing | 7

52. Secondary Outcome: Knee Function and Stability: Extension Stability at 52 Weeks
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: 52 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 22
  Abnormal instability | 1
  Instability in extension <10 degrees | 1
  Instability in extension >10 degrees | 0
  Missing | 4

53. Secondary Outcome: Knee Function and Stability: Extension Stability at 78 Weeks
Description: Knee extension stability was evaluated by the investigator right after surgery (Baseline) and at each follow-up visit.
Time Frame: 78 weeks
Population: Five major protocol violations were excluded in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 28
participants
  Normal stability | 17
  Abnormal instability | 3
  Instability in extension <10 degrees | 1
  Instability in extension >10 degrees | 0
  Missing | 7

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline (surgery) through the end of the follow-up period at 78 or 104 weeks (Australian sites only).
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 15/33
Other Adverse Events (participants affected / at risk) | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=33)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1)
DEVICE EXTRUSION (General disorders) | 1 (1)
INFLAMMATION (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
HEPATIC CIRRHOSIS (General disorders) | 1 (1)
INFECTION (Infections and infestations) | 2 (2)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
LOSS OF ANATOMICAL ALIGNMENT AFTER FRACTURE REDUCTION (Injury, poisoning and procedural complications) | 2 (2)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
TENDON PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=33)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
MEDICAL DEVICE PAIN (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
DEVICE EXTRUSION (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
LOSS OF ANATOMICAL ALIGNMENT AFTER FRACTURE REDUCTION (Injury, poisoning and procedural complications) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
FRACTURE DELAYED UNION (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1)
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less